CLINICAL TRIAL: NCT06366763
Title: Comparative Clinical Efficacy Between Multi-layer Bandage Pressure Therapy and Compression Stockings Treatment After Endovenous Radiofrequency Ablation
Brief Title: Comparative Clinical Efficacy Between Multi-layer Bandage Pressure Therapy and Gradient Pressure Elastic Stocking Treatment After Endovenous Radiofrequency Ablation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunshui He, chief physician, Chengdu University of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChengduUTCMvs5
Record Dates: First submitted 2024-01-20; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Vascular Diseases, Peripheral; Venous Insufficiency of Leg; Varicose Veins of Lower Limb
Keywords: Gradient pressure elastic stockings; Varicose veins; Radiofrequency ablation; Compression therapy
MeSH Terms: conditions — Peripheral Vascular Diseases; Varicose Veins | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Among the 210 patients included in the study (82 males, 128 females; average age of 59 years), 7 patients were lost to follow-up, and the remaining patients completed the treatment and follow-up.To assess the clinical efficacy of different compression methods within 48 hours after endovenous radiofrequency ablation (RFA) in terms of great saphenous vein closure rate, postoperative complications, quality of life, time to return to normal work, and patient satisfaction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gradient pressure elastic stocking treatment after endovenous radiofrequency ablation. (Experimental): Among the 210 patients to assess the clinical efficacy of different compression methods within 48 hours after endovenous radiofrequency ablation (RFA) in terms of great saphenous vein closure rate, postoperative complications, quality of life, time to return to normal work, and patient satisfaction.
  Interventions: Procedure: Questionnaires

INTERVENTIONS:
Procedure: Questionnaires — Questionnaires to assess the quality of life (CIVIQ-14 and VCSS scores )

SUMMARY:
Objective: To assess the clinical efficacy of different compression methods within 48 hours after endovenous radiofrequency ablation (RFA) in terms of great saphenous vein closure rate, postoperative complications, quality of life, time to return to normal work, and patient satisfaction.

DETAILED DESCRIPTION:
Postoperative compression of varicose veins can achieve compression hemostasis, early getting out of bed, reducing edema, preventing phlebitis, ensuring closure effect, reducing soreness and pain, and preventing thrombosis. Compression therapy is a continuation of minimally invasive treatment of varicose veins, and postoperative compression therapy is continued for at least 1 month, and grade II compression therapy may be considered.The application of postoperative compression to the treated limb after radiofrequency ablation of the great saphenous vein has been a topic of controversy. The basic principle of using postoperative compression is to reduce the risk of bleeding, hematoma formation, pain, swelling, and thrombus formation. However, many patients find wearing gradient pressure elastic stockings cumbersome and uncomfortable, as the silicone grips around the stockings can cause skin itching and discomfort. Moreover, there is a lack of strong evidence supporting this treatment. The purpose of this study was to investigate the effectiveness of continuous 48-hour use of gradient pressure elastic stockings for compression of the affected limb after endovenous radiofrequency ablation.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years and <80 years, and able to understand the requirements of the study and provide informed consent and accept the exams and follow-up.
* C2 - C5 varicose veins / CVI Symptomatic primary GSV, SSV, or AASV incompetence, with reflux >0.5 seconds on color duplex, eligible for patients undergoing radiofrequency ablation.
* Color replica ultrasound or venography of the lower extremity veins shows saphenous varicose veins without evidence of deep venous stenosis, filling defects, or ultrasound abnormalities.
* No contraindications to the wearing of compression stockings (e.g., arterial insufficiency, skin allergies)

Exclusion Criteria:

* Severe deep vein valve insufficiency or acute deep vein thrombosis of the lower extremities
* Previous history of high ligation and dissection of the saphenous vein, recurrence of collateral branches of the deep vein
* Superficial vein thrombosis is present at the treatment site, with local redness, swelling, warmth, pain, and significant signs of inflammation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain after radiofrequency ablation | 2 days post-procedure
  Pain is assessed using a visual analogue score (1-10), with higher scores representing more pronounced pain。
Bleeding after radiofrequency ablation | 2 days post-procedure
  Through the observation of ward rounds and telephone follow-up of patients in the hospital, the frequency of postoperative lower limb bleeding events was obtained, with 0 representing no bleeding events and 1 representing bleeding events
Tension blisters after radiofrequency ablation | 2 days post-procedure
  Through the observation of ward rounds and telephone follow-up of patients in the hospital, the frequency of postoperative lower extremity skin tension blister events was obtained, with 0 indicating negative and 1 indicating positive

SECONDARY OUTCOMES:
The rate of occlusion of treated vein post-procedure | 2 days, 1 month, 3 months, 1 year after surgery
  Use duplex ultrasound assess the occlusion of treated vein post-procedure,record the rate of occlusion of treated vein post-procedure
Quality of life score using the Chronic Venous Insufficiency Questionnaire(CIVIQ-14) | 2 days, 1 month, 3 months, 1 year after surgery
  CIVIQ-14 is a questionnaire based on three dimensions - pain, physical and psychological, based on a scale from 1 to 5 (no trouble, slight, moderate, considerable, severe).Based on inputs, CIVIQ-14 will be tabulated, ranging from 0 to 100 - the higher the value, the poorer the quality of life.In order to observe the changes in quality of life over the whole test procedure.
Clinical Change using Venous Clinical Severity Score (VCSS) | 2 days, 1 month, 3 months, 1 year after surgery
  VCSS evaluates the severity of hallmarks of venous disease - 0 (none), 1 (Mild) , 2(Moderate), 3 (Severe).Record the score separately to observe the changes in quality of life over the whole test procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Epstein D, Bootun R, Diop M, Ortega-Ortega M, Lane TRA, Davies AH. Cost-effectiveness analysis of current varicose veins treatments. J Vasc Surg Venous Lymphat Disord. 2022 Mar;10(2):504-513.e7. doi: 10.1016/j.jvsv.2021.05.014. Epub 2021 Aug 25. PMID 34450353
- [Result] Karathanos C, Spanos K, Batzalexis K, Nana P, Kouvelos G, Rousas N, Giannoukas AD. Prospective comparative study of different endovenous thermal ablation systems for treatment of great saphenous vein reflux. J Vasc Surg Venous Lymphat Disord. 2021 May;9(3):660-668. doi: 10.1016/j.jvsv.2020.10.008. Epub 2020 Oct 21. PMID 33099037
- [Result] Siribumrungwong B, Noorit P, Wilasrusmee C, Attia J, Thakkinstian A. A systematic review and meta-analysis of randomised controlled trials comparing endovenous ablation and surgical intervention in patients with varicose vein. Eur J Vasc Endovasc Surg. 2012 Aug;44(2):214-23. doi: 10.1016/j.ejvs.2012.05.017. Epub 2012 Jun 15. PMID 22705163
- [Result] Poder TG, Fisette JF, Bedard SK, Despatis MA. Is radiofrequency ablation of varicose veins a valuable option? A systematic review of the literature with a cost analysis. Can J Surg. 2018 Apr;61(2):128-138. doi: 10.1503/cjs.010114. PMID 29582749
- [Result] Lawaetz M, Serup J, Lawaetz B, Bjoern L, Blemings A, Eklof B, Rasmussen L. Comparison of endovenous ablation techniques, foam sclerotherapy and surgical stripping for great saphenous varicose veins. Extended 5-year follow-up of a RCT. Int Angiol. 2017 Jun;36(3):281-288. doi: 10.23736/S0392-9590.17.03827-5. Epub 2017 Feb 17. PMID 28217989
- [Result] Staubesand J, Seydewitz V. [An ultrastructural study of sclerosed varices]. Phlebologie. 1991 Jan-Mar;44(1):16-22; discussion 33-6. French. PMID 1946638
- [Result] Lurie F, Lal BK, Antignani PL, Blebea J, Bush R, Caprini J, Davies A, Forrestal M, Jacobowitz G, Kalodiki E, Killewich L, Lohr J, Ma H, Mosti G, Partsch H, Rooke T, Wakefield T. Compression therapy after invasive treatment of superficial veins of the lower extremities: Clinical practice guidelines of the American Venous Forum, Society for Vascular Surgery, American College of Phlebology, Society for Vascular Medicine, and International Union of Phlebology. J Vasc Surg Venous Lymphat Disord. 2019 Jan;7(1):17-28. doi: 10.1016/j.jvsv.2018.10.002. PMID 30554745